CLINICAL TRIAL: NCT02099461
Title: A Randomized, Stratified, Open-label, No-treatment-controlled, Parallel Group, Multicenter Phase 1 Trial to Evaluate the Effect of Denosumab on Cellular Proliferation in the Human Breast
Brief Title: Effect of Denosumab on Cellular Biomarkers in the Human Breast
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20130349
Record Dates: First submitted 2014-02-25; First posted 2014-03-31 (Estimated); Results first posted 2015-09-24 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-08

CONDITIONS: Healthy Volunteer, Female, Breast
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No treatment (Other): Participants received no treatment and underwent percutaneous core needle breast biopsies on Day 1 and Day 28.
  Interventions: Procedure: Percutaneous core needle breast biopsy
- Denosumab 60 mg (Experimental): Participants received 60 mg denosumab by subcutaneous injection on Day 1 and underwent percutaneous core needle breast biopsies on Day 1 (prior to study treatment) and Day 28.
  Interventions: Drug: Denosumab; Procedure: Percutaneous core needle breast biopsy
- Denosumab 120 mg (Experimental): Participants received 120 mg denosumab by subcutaneous injection on Day 1 and underwent percutaneous core needle breast biopsies on Day 1 (prior to study treatment) and Day 28.
  Interventions: Drug: Denosumab; Procedure: Percutaneous core needle breast biopsy

INTERVENTIONS:
Drug: Denosumab — Single sucutaneous dose
  Arms: Denosumab 120 mg; Denosumab 60 mg
Procedure: Percutaneous core needle breast biopsy

SUMMARY:
To evaluate whether administration of denosumab results in a decrease compared to the control group in proliferation of mammary epithelial cells as measured by the Ki-67 proliferation index.

ELIGIBILITY:
INCLUSION CRITERIA:

* Willing to use, in combination with her partner, 2 non-hormonal methods of effective contraception or practice sexual abstinence. Subjects who are surgically sterile (eg, history of hysterectomy) or whose sexual partner is sterile (eg, history of vasectomy) are not required to use contraceptive measures
* Laboratory tests are within clinically acceptable range
* Clinically acceptable physical exam and no history or evidence of any clinically significant medical disorder that would pose a risk to subject safety or interfere with study evaluations or procedures.

EXCLUSION CRITERIA:

* Female subject with a prior history of breast cancer; breast implant in the breast to be biopsied; Known history of fibrocystic breast disease
* Subject is unable or unwilling to provide breast biopsy tissue from the upper outer quadrant of her breast
* Pregnant or plans to become pregnant while exposed to investigational product
* Lactating/breastfeeding or plans to breastfeed while exposed to investigational product
* Recent use of any non-approved medications or devices
* Uncontrolled thyroid disorder
* Significant dental/oral disease
* Planned invasive dental procedures
* Positive urine screen for alcohol and/or drugs

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- United States (3):
  - Research Site, Cypress, California
  - Research Site, Hollywood, Florida
  - Research Site, Miami, Florida

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: On study day 1, eligible participants were randomized into 1 of 3 treatment assignments. Randomization was stratified by average length of menstrual cycle (< 28 days, equal to 28 days, and > 28 days).
Groups:
- Denosumab 60 mg: Participants received 60 mg denosumab by subcutaneous injection on Day 1 and underwent percutaneous core needle breast biopsies on Day 1 and Day 28.
- Denosumab 120 mg: Participants received 120 mg denosumab by subcutaneous injection on Day 1 and underwent percutaneous core needle breast biopsies on Day 1 and Day 28.
Period: Overall Study
Arm/Group | No Treatment | Denosumab 60 mg | Denosumab 120 mg
Started | 27 | 27 | 28
Completed | 27 | 27 | 28
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Treatment | Denosumab 60 mg | Denosumab 120 mg | Total
Number analyzed (Participants) | 27 | 27 | 28 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.9 (7.3) | 32.2 (7.6) | 32.8 (8.8) | 32.5 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 28 | 82
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 0 | 1 | 1
  Black (or African American) | 4 | 8 | 10 | 22
  Multiple | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2
  Whte | 21 | 19 | 16 | 56

OUTCOME MEASURES:

1. Primary Outcome: Log Ratio of Post-baseline to Baseline Ki-67 Index in Mammary Epithelial Cells
Description: Ki-67 is a marker for cell proliferation. Participants underwent percutaneous core needle breast biopsies on Day 1 (Baseline, prior to treatment) and Day 28. Levels of Ki67 were measured using immunohistochemical staining and digital imaging. The proliferation index was calculated as the percentage of Ki-67 positive terminal ductal lobular unit (TDLU) and duct epithelial cells. The higher the percentage, the higher the rate of epithelial cell proliferation.
Time Frame: Baseline and Day 28
Population: Pharmacodynamic analysis set with non-missing data
Measure: Mean (Standard Deviation); unit: log ratio
Arm/Group | No Treatment | Denosumab 60 mg | Denosumab 120 mg
Number analyzed (Participants) | 25 | 25 | 26
log ratio | 0.084 (0.645) | -0.100 (1.048) | -0.081 (0.918)
Statistical Analysis 1: Comparison: No Treatment; An ANCOVA analysis was performed on the log ratio of post-baseline to baseline Ki-67 index. Independent variables included treatment, stratification factor, and log transformed baseline Ki-67 index; Test type: Superiority or Other; p = 0.2966, ANCOVA; LS Mean = 0.15, 95% CI 2-sided [-0.136 to 0.441]
Statistical Analysis 2: Comparison: Denosumab 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2769, ANCOVA; LS Mean = -0.16, 95% CI 2-sided [-0.447 to 0.130]
Statistical Analysis 3: Comparison: Denosumab 120 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5238, ANCOVA; LS Mean = -0.09, 95% CI 2-sided [-0.373 to 0.191]
Statistical Analysis 4: Comparison: No Treatment vs Denosumab 60 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1343, ANCOVA; LS Mean Difference = -0.31, 95% CI 2-sided [-0.720 to 0.098] — Denosumab 60 mg - Placebo
Statistical Analysis 5: Comparison: No Treatment vs Denosumab 120 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.2345, ANCOVA; LS Mean Difference = -0.24, 95% CI 2-sided [-0.646 to 0.161] — Denosumab 120 mg - Placebo

ADVERSE EVENTS:
Time Frame: 28 days
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Treatment A No Treatment: Participants in this group received no treatment and underwent percutaneous core needle breast biopsies on Day 1 and Day 28.
- Treatment B 60 MG SC: Participants received 60 mg denosumab by subcutaneous injection on Day 1 and underwent percutaneous core needle breast biopsies on Day 1 and Day 28.
- Treatment C 120 MG SC: Participants received 120 mg denosumab by subcutaneous injection on Day 1 and underwent percutaneous core needle breast biopsies on Day 1 and Day 28.
Arm/Group | Treatment A No Treatment | Treatment B 60 MG SC | Treatment C 120 MG SC
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 4/27 | 6/27 | 11/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A No Treatment (N=27) | Treatment B 60 MG SC (N=27) | Treatment C 120 MG SC (N=28)
Injection site erythema (General disorders) | 0 | 1 | 10
Procedural pain (Injury, poisoning and procedural complications) | 4 | 4 | 2
Headache (Nervous system disorders) | 0 | 0 | 2
Breast haematoma (Reproductive system and breast disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.